CLINICAL TRIAL: NCT07144852
Title: Randomized, Multi-Center, Evaluator-Blind, Vehicle-Controlled Study to Evaluate Efficacy and Safety of Reformulated Levulan Kerastick Plus Photodynamic Therapy (PDT) for Field-Directed Treatment in Patients With Actinic Keratosis (AK) of Upper Extremities
Brief Title: Study of Reformulated Levulan Kerastick Plus PDT for Actinic Keratosis on Upper Extremities
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Organization: Sun Pharmaceutical Industries Limited (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LEV-24-01
Record Dates: First submitted 2025-08-20; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Actinic Keratosis
Keywords: Blue Light Photodynamic Therapy, Skin Diseases, Precancerous Conditions, Photosensitizing Agents, Dermatologic Agents, Aminolevulinic Acid
MeSH Terms: conditions — Keratosis, Actinic; Skin Diseases; Precancerous Conditions | interventions — Aminolevulinic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participant, investigator and outcomes assessor are blinded to treatment assignment, as both Levulan and Vehicle products look identical and cannot be differentiated from the application characteristics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Levulan (Experimental): Levulan application + incubation time (with occlusion) + blue light application
  Interventions: Drug: Reformulated Levulan Kerastick containing aminolevulinic acid hydrochloride (ALA HCl), 20%; Device: Blue Light Photodynamic Therapy Illuminator device, BLU-U® model 4170E.
- Vehicle (Placebo Comparator): Vehicle application + incubation time (with occlusion) + blue light application
  Interventions: Other: Vehicle; Device: Blue Light Photodynamic Therapy Illuminator device, BLU-U® model 4170E.

INTERVENTIONS:
Drug: Reformulated Levulan Kerastick containing aminolevulinic acid hydrochloride (ALA HCl), 20% — Solution for topical use
  Arms: Levulan
Other: Vehicle — Solution for topical use
  Arms: Vehicle
Device: Blue Light Photodynamic Therapy Illuminator device, BLU-U® model 4170E. — BLU-U® blue light PDT illuminator

SUMMARY:
This Phase 3, randomized, multi-center, evaluator-blind, vehicle-controlled study evaluates the efficacy and safety of reformulated Levulan Kerastick (aminolevulinic acid HCl 20%) combined with photodynamic therapy (PDT) for field-directed treatment of actinic keratosis (AK) on the upper extremities. Approximately 260 adult patients with 4-8 mild to moderate AK lesions on one arm will be randomized to receive either active treatment or vehicle control, followed by exposure to blue light. During the study, up to 2 PDT sessions may be administered depending on the clearance of lesions. The primary endpoint is complete clearance rate (CCR) at Week 12. Secondary endpoints include AK clearance rate (AKCR), partial clearance, change in total lesion count and area, recurrence rate, cosmetic response, and patient satisfaction. Safety assessments include adverse events, local skin reactions, vital signs, and lab tests.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is a male or non-pregnant female aged 18-85 years.
2. Patient must have 4-8 mild to moderate actinic keratosis (AK) lesions (Olsen grade 1 or 2) in a single treatment area on their Index arm, each measuring up to 1 cm in diameter and spaced at least 1 cm apart.

   [The treatment area should be approximately 25 cm², located on the extensor surface of only one of the upper extremities that is selected as the Index arm]
3. Patients must be in good general health, avoid sunbathing or tanning devices, and maintain a consistent skincare routine throughout the study.
4. Patient is willing to stop using all topical products within the Treatment Area within 8 hours of a scheduled clinic visit with an efficacy evaluation.
5. Women of childbearing potential must use highly effective contraception; men with such partners must use barrier methods unless surgically sterile.

Exclusion Criteria:

1. Presence of Olsen grade 3 AK, untreated or suspicious skin cancers, or significant skin abnormalities (e.g., psoriasis, eczema) in the treatment area.
2. Active herpes simplex infection or history of ≥2 outbreaks in the treatment area within the past year.
3. History of cutaneous photosensitization, porphyria, photodermatosis, or hypersensitivity to porphyrins.
4. Positive human immunodeficiency virus (HIV) test result, hepatitis B surface (HBS) antigen, or hepatitis C virus (HCV) test result
5. Immunosuppressed status (e.g., HIV, organ transplant) or known coagulation defects.
6. Use of specific topical therapies (e.g., retinoids, steroids, cryotherapy, PDT, chemical peels) on the treatment area within 2 days to 8 weeks prior to randomization.
7. Recent use of certain systemic therapies (e.g., corticosteroids, immune-modulators, retinoids, cytotoxic drugs) within 6 weeks to 6 months prior to randomization.
8. Recent use of hypericin or other phototoxic/photoallergic medications (e.g., tetracyclines, psoralenes, St. John's wort) within 8 weeks of randomization.
9. Clinically significant or unstable illnesses, or history of alcohol/drug abuse in the past year.
10. Pregnancy/lactation, recent or current participation in another clinical study, or any other condition deemed unsuitable by the Investigator.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-06-29 (Estimated); Study Completion 2026-09-24 (Estimated)

PRIMARY OUTCOMES:
Complete Clearance Rate (CCR) i.e., proportion of patients achieving complete clearance of all AK lesions in the Treatment Area) | Week 12
  Complete clearance is defined as clearance of all AK lesions in the Treatment Area after PDT 1 or PDT 2, if re-treated; lesions should no longer be palpable nor visible to be declared as "cleared"

SECONDARY OUTCOMES:
Actinic Keratosis Clearance rate (AKCR) | Week 4, 8 ,12, 20, and 24
  AKCR for each patient is calculated as 100 x [1- (number of target AK lesions present at that particular visit/ number of target AK lesions present at Baseline)]. Target lesions are those AK lesions that were identified at baseline and treated at baseline
Proportion of patients achieving clearance of target lesions in the Treatment Area | Weeks 4, 8, 12, 20, and 24
  Target lesions are those AK lesions that were identified at baseline and treated at baseline.
Complete Clearance Rate (CCR) i.e., proportion of patients achieving complete clearance of all AK lesions in the Treatment Area | Weeks 4, 8, 20, and 24
Partial Clearance Rate (PCR); i.e., Proportion of patients achieving partial clearance of AK lesions) | Weeks 4, 8, 12, 20, and 24
  Partial clearance is defined as clearance of at least 75% of all AK lesions in the Treatment Area; lesions should no longer be palpable nor visible to be declared as "cleared".
Percent change in total AK lesion count from Baseline | Weeks 4, 8, 12, 20, and 24
Percent change in total AK lesion area from Baseline | Weeks 8, 12, and 24
Investigator Assessment of Cosmetic Response | Weeks 12, 20, and 24
  The overall cosmetic response to treatment will be assessed by a Blinded Investigator using a 4-point scale, selecting the score that best describes the patient's cosmetic outcome in actinic keratosis since treatment initiation: 1 = Excellent, 2 = Good, 3 = Fair, and 4 = Poor.
Patient Assessment of Cosmetic Response | Weeks 12, 20, and 24
  The patient's overall cosmetic response to treatment will be measured by the patient on a 4-point scale, where 1 = Excellent, 2 = Good, 3 = Fair, and 4 = Poor
Patient Satisfaction Score (PSS) at Weeks 12, 20, and 24. | Weeks 12, 20, and 24
  The patient's overall satisfaction with the study treatment will be assessed using a 4-point patient-reported scale, where 0 = Not satisfied at all, 1 = Slightly satisfied, 2 = Moderately satisfied, and 3 = Very satisfied.
Recurrence Rate at Week 24. Measured as proportion of patients presenting with at least one recurrent lesion during the follow-up period, after having achieved complete clearance at Week 12. | Week 24
  Measured as proportion of patients presenting with at least one recurrent lesion during the follow-up period, after having achieved complete clearance at Week 12.